CLINICAL TRIAL: NCT02933424
Title: The Effects of Plant Proteins on Blood Glucose & Amino Acid Levels and Satiety in Humans
Brief Title: Project Plant Protein: the P3 Study in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016/00796
Record Dates: First submitted 2016-09-27; First posted 2016-10-14 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Pre-diabetes; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control beverage with no protein powder (No Intervention): Standard breakfast drink with no protein powder added
- Beverage with Rice protein powder 25 grams (Experimental): Standard breakfast drink with 25 grams of rice protein powder.
  Interventions: Dietary Supplement: Protein Powder
- Beverage with Pea protein powder 25 grams (Experimental): Standard breakfast drink with 25 grams of pea protein powder.
  Interventions: Dietary Supplement: Protein Powder
- Beverage with Oats protein powder 25 grams (Experimental): Standard breakfast drink with 25 grams of Oats protein powder.
  Interventions: Dietary Supplement: Protein Powder

INTERVENTIONS:
Dietary Supplement: Protein Powder
  Arms: Beverage with Oats protein powder 25 grams; Beverage with Pea protein powder 25 grams; Beverage with Rice protein powder 25 grams

SUMMARY:
The objective of this study is to compare the effects of adding three plant-based proteins (rice, oats and pea proteins) to a breakfast beverage on the glycemic response, appetite and subsequent food intake of healthy adults.

DETAILED DESCRIPTION:
A diet or a meal higher in dietary protein has been reported to promote satiety and suppress food intake in humans in several previous studies. It was suggested that the presence of amino acid in the blood as a result of higher protein intake served as signals that suppress appetite in humans. More recently, it has been observed that incomplete or lower quality proteins, i.e. those missing one or more essential amino acids, may suppress hunger more than complete proteins, as the ingestion of incomplete proteins in the long term may lead to deficiency of essential amino acids. Plant proteins are generally considered incomplete protein when compared to animal proteins, which mean that plant protein may have higher appetite-suppressing effects.

Dietary carbohydrates are the most potent stimuli of insulin secretion. However, the addition of dietary protein in a carbohydrate-rich meal has been shown to further stimulate insulin release.The insulinotropic effect of dietary protein is thought to be attributed to the branched-chain amino acid (BCAA) content of the protein-rich meal. Interestingly, there is a hierarchy of effects induced by protein from different sources. For example, milk protein has been shown to be superior to fish or plant protein in stimulating insulin secretion following a meal.Even within milk protein, whey protein stimulated insulin secretion more than casein protein. One of the factors that distinguish whey from casein proteins was the digestibility or the digestion rate of these proteins. Protein that is digested faster appear to increase blood amino acid levels faster, and increase insulin release faster.This implies that plant proteins that have lower digestibility rate relative to animal proteins may have lower insulinotropic effects, and the effective dose required to achieve optimal insulin secretion may be different from animal protein and warrants further investigation. In addition, the amino acid profile (in addition to lower digestibility) of plant proteins may differ from animal protein, especially the BCAA content that is associated with the stimulation of insulin secretion.

Dietary patterns and cuisines vary between countries and cultures. Unlike in the Western countries, plant-based foods are more commonly consumed in an Asian cuisine. Based on the statistics released by Food and Agriculture Organization, cereals and meat are the top two protein sources in both Western (29.1% and 26.4% respectively) and Asian (58.8% and 8.6% respectively) countries. The third major source of protein is dairy (16.7%) in Western countries, and pulses in Asia (7.4%). In addition, vegetarianism is widely practiced in Asian countries. Studies investigating the appetitive and the blood glucose regulating effects of dietary protein have been focused predominantly in animal protein, with a number of studies included plant-based protein such as soy protein. Since cereals and pulses are an important part of an Asian cuisine, it is important to understand and compare the effects of proteins from these sources on blood glucose and appetite regulation. Since the amino acid profile and the digestibility of these plant-based proteins differ from animal protein, it is important to also understand the effective dose that exerts optimal effects.

ELIGIBILITY:
Inclusion Criteria:

* Males
* BMI 18.5-24.9kgm-2
* eating all meals (5 days/week)

Exclusion Criteria:

* major chronic disease such as heart disease, cancer, hypertension or diabetes mellitus
* have gout
* have food allergies
* are taking insulin or drugs known to affect metabolism, appetite and body fat distribution,
* have weight change of >5kg in the past 3 months
* have major medical or surgical event requiring hospitalisation within the preceding three months
* are on a weight loss regime, and presence of disease or drugs which influence digestion and absorption of nutrients
* smokers,
* individuals who take part in sports at competitive/endurance levels

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose | Up to 180 minutes
  Blood glucose measured up to 180 minutes
Change in blood insulin | Up to 180 minutes
  Blood insulin measured up to 180 minutes
Change in gut hormones | Up to 180 minutes
  Blood gut hormones measured up to 180 minutes
Change in body weight | At baseline
  Body weight measured with a Bio-electrical impedance scale
Change in body composition | At baseline
  Fat% measured with a Bio-electrical impedance scale

SECONDARY OUTCOMES:
Change in subjective appetite ratings | Up to 180 minutes
  Appetite ratings measured up to 180 minutes
Change in plasma amino acid | Up to 180 minutes
  Blood amino acid profile measured up to 180 minutes
Meal challenge | At 180 minutes
  Ad libitum meal challenge at 180-minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

REFERENCES:
- [Derived] Tan SY, Siow PC, Peh E, Henry CJ. Influence of rice, pea and oat proteins in attenuating glycemic response of sugar-sweetened beverages. Eur J Nutr. 2018 Dec;57(8):2795-2803. doi: 10.1007/s00394-017-1547-3. Epub 2017 Sep 30. PMID 28965176